CLINICAL TRIAL: NCT04272268
Title: Evaluating the Feasibility and Safety of Using Nasal High Flow Oxygen for Five Days Postoperatively to Reduce Respiratory Complications After Oesophagectomy for Cancer
Brief Title: Feasibility and Safety of Using Nasal High Flow Oxygen Postoperatively to Reduce Respiratory Complications
Acronym: Hi-FLO
Status: Withdrawn | Type: Observational
Why Stopped: Covid-19
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2063; 214643 (Other: IRAS)
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-12

CONDITIONS: Cancer of the Esophagus
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nasal High flow Oxygen: Following consent, the participant will undergo Oesophagectomy as per routine care. During surgery, prior to trial participation and as per standard of care at the site, a nasogastric tube will be placed into the gastric conduit and secured to the nose. This tube will be left on free drainage and aspirated every 4 hours to check for inadvertent insufflation.
  Interventions: Device: Nasal High flow Oxygen

INTERVENTIONS:
Device: Nasal High flow Oxygen — If the patient is successfully extubated within 4 hours following surgery and meets the post surgery inclusion/exclusion criteria, Nasal high flow oxygen will be administered continuously using a humidifier machine for 5 days. Breathing circuits and nasal cannulae will be connected to the machine to deliver oxygen at 20L/min to the patient.

SUMMARY:
The use of nasal high flow in patients undergoing oesophagectomy is a novel technique that has not been previously studied.

Nasal high flow will be delivered postoperatively to patients undergoing oesophagectomy in a tertiary cancer referral centre. This single-centre cohort study will evaluate the safety of using nasal high flow in oesophagectomy patients. Physiological parameters, adverse events and clinical outcome will be recorded in consecutive patients undergoing oesophagogastric surgery.

This study will challenge the hypothesis that the use of nasal high-flow will lower the rates of breathing complications such as pneumonia thereby reducing the demands on intensive care, shortening hospital stay and improving patient quality of life. The results will inform the design of a larger multicentre clinical trial comparing nasal high flow to conventional methods by facilitating sample size calculation.

DETAILED DESCRIPTION:
Respiratory complications including pneumonia, pleural effusion, adult respiratory distress syndrome and pulmonary embolism will be recorded. The primary endpoint will be the rate of postoperative respiratory complications within 30 days of oesophagectomy. Technical complications related to nasal high flow administration will be recorded and reasons for discontinuing nasal high flow documented. Other outcome including mortality, hospital stay, surgical complications and respiratory complications within 90 days of surgery will be considered as secondary endpoints. These data will assess the feasibility and safety of using nasal high flow in patients undergoing oesophagectomy. The rate of respiratory complications will be determined in a cohort of consecutive surgical patients together with other measures of outcome to form the basis of a series worthy of reporting. This may help gain insight into whether using nasal high flow could benefit patients, and whether further research to compare nasal high flow to conventional respiratory support would be of value.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Undergoing Ivor-Lewis (2-stage) oesophagectomy
* Successfully extubated within 4 hours after surgery

Exclusion Criteria:

* History of bullous emphysematous disease
* Lack of capacity to consent
* Significant air leak during surgery
* Incurable disease found at surgery leading to no surgical resection
* Failure of extubation and spontaneous breathing within 4 hours after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nasal high flow will be delivered postoperatively to patients undergoing oesophagectomy in a tertiary cancer referral centre. This single-centre cohort study will evaluate the safety of using nasal high flow in oesophagectomy patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of respiratory complications within 30 days after surgery | 30 days
  including pneumonia, pleural effusion, adult respiratory distress syndrome and pulmonary embolism.

SECONDARY OUTCOMES:
30 day mortality | 30 days
90 day mortality | 90 days
90 day respiratory complication rate | 90 days
The proportion of blood gases performed on time | 5 days
The proportion of missing results | 5 days
Recruitment rate | 90 days
  To facilitate sample size calculation for such a randomized controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Gerorge Bouras, Principal Investigator — University Hospitals of North Midlands NHS Trust
Locations (1):
- Robert James Bowler, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No